CLINICAL TRIAL: NCT06370650
Title: Effect of Platelet Rich Plasma on Outcome of Narrow Band UVB in Treatment of Vitiligo; Clinical and Histopathological Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Hassan Ahmed, assissant lecturer, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-24-1-9
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Management of Stable Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrow band UVB (Active Comparator)
  Interventions: Procedure: platelet rich plasma, narrow band UVB
- Platelet rich plasma plus narrow band UVB (Active Comparator)
  Interventions: Procedure: platelet rich plasma, narrow band UVB

INTERVENTIONS:
Procedure: platelet rich plasma, narrow band UVB — Role of PRP in treating stable vitiligo

SUMMARY:
For each patient, one side of body will be treated with NB-UVB alone while the other side will be treated with NB-UVB therapy in addition to intradermal injection of PRP every 2 weeks. Patients will be photographed at the first visit, in the middle and at the end of therapy. Each patient will sign a written consent form to be included in the study and to be photographed.

ELIGIBILITY:
Inclusion Criteria:

Patients with stable non segmental vitiligo. (Absence of koebnerization, absence of new lesion and absence of widening of the existing lesions).

Patients have more than 15 years.

-

Exclusion Criteria:

Patients have active vitiligo (appearance of new lesion, history of koebnerization).

Pregnant and lactating women. History of keloid formation. Anemia (hemoglobin level <10gm/dl), thrombocytopenia (platelet count <100,000 /µL), coagulopathies or patients on anticoagulant therapy and patients with iron deficiency.

Patients taking drugs that prolong bleeding time such as Aspirin and vitamin E Patients taking treatment of vitiligo in last 2 months

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of vitiligo | within 6 months
  increase repigmentation score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Researcher shall pubish in national journal